CLINICAL TRIAL: NCT06034171
Title: Clinical Study of Implants With Modified Surface Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SmileDent Kft. (Industry)
Collaborators: S.G.S International Kft. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SM-SGS_001
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Dental Implant; Hydroxyapatite
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Intervention Model Description: two arms, split-mouth, randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (study implant on the right side) (Experimental): Implant with phosphate surface device in the right side of the lower jawbone, and the hydroxylapatite surface treatment implant is placed in the left side of the lower jaw.
  Interventions: Device: dental implant
- Group B (study implant on the left side) (Experimental): Implant with phosphate surface device for the lower jaw on the left side, and the implant with hydroxylapatite surface treatment is inserted into the right side of the jawbone.
  Interventions: Device: dental implant

INTERVENTIONS:
Device: dental implant — Dental implant surgery in the lower jawbone.

SUMMARY:
The observed medical device in this study were SGS P7D Dental implant. The device replaces the lost tooth root, and provides support for the dental bridges and crowns, or overdenture replacements. This medical device provides the opportunity to to replace partial or complete missing teeth. Device material: Ti-6Al-4V Device surface protection: Corundum Blasting and

1. phosphate surface treatment or
2. hydroxylapatite surface treatment

DETAILED DESCRIPTION:
A prospective, randomized, two-arms "split-mouth" study. The two arms: right and left of the same mandible of the same volunteer with a different surface treatment, but every other circumstances of the implants are the same, the same device with different surface materilas.

"A" treatment: Implant with phosphate surface treatment is the lower one in the right side of the jawbone, with hydroxylapatite surface treatment implant is placed in the left side of the lower jaw. "B" treatment: Implant with phosphate surface treatment in the lower jaw on the left side, the bottom is an implant with hydroxylapatite surface treatment is inserted into the right side of the jaw bone

ELIGIBILITY:
Inclusion Criteria:

* complete lack of teeth in the lower jaw
* decision of the investigator: the patient is appropriate for implantation, clinical conditions are sufficient (adequate soft tissue and bone conditions and occlusal position;)
* the patient's consciousness is clear, understand the planned intervention.
* the patient communicates well with the examiner and is able to understand and comply with the requirements of the test plan.
* witten informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Women of childbearing potential, unless she uses effective birth control until the completion of the final radiological examination, and for another 4 weeks after that.
* A disease (including, but not limited to metabolic, hematological, kidney, liver, lung, neurological, endocrine, cardiac, infectious and gastrointestinal disease), which -in the opinion of the investigator- significantly affects the health of the examined person and/or exposes to an unacceptably high risk the person receiving the implantation treatment.
* Malignant disease in the medical history in the preceding 24 months.
* Known HIV, hepatitis B or hepatitis C, or any other considered viral infection relevant by the examiner known at the tome of randomization
* A medical or psychiatric illness which, in the opinion of the investigator, excludes that the participant adheres to the protocol, or complete the study according to the protocol.
* Participation in an other interventional clinical study within 6 months prior to treatment.
* Known allergy to the implant or to the invetigational template or any of its components.
* Limitation of mouth opening, which make unpossible to complete the procedure, based on the opinion of the investigator
* Increased pharyngeal reflex, reduced ability to tolerate intraoral manipulation
* Radiotherapy, previous irradiation of the jawbones
* INR > 2.5
* Immunosuppressed patient
* previous or current bisphosphonate treatment
* Known alcohol or drug abuse
* Heavy smoking (≥ 20 cigarettes per day, or another form of smoking, used in an equivalent amount)
* Untreated periodontitis
* Local infection of the implant in the planned area
* Lack of dental hygiene, e.g. not removed radixes, plaque and calculus, or radiologically detectable potential periapical focus (also in asymptomatic case )
* Insufficient or poor oral hygiene
* Transient infectious state, with or without fever

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of OSSTELL ISQ score (for the degree of osseointegration indicator) | 36 months
  Evaluation the difference between the two types surface treated implants osseointegration. For the measure is used the OSSTELL ISQ score.
  results with the OSSTELL radio frequency device based on measurable stability values. Values can vary form 1-100, higher values mean better stability.

SECONDARY OUTCOMES:
Volunteer-Quality of Life (OHIP Scale Scores) | 36 months
  Establishing the effect of implantation and subsequent prosthetic intervention on the volunteers long-term quality of life based on the scales of the OHIP questionnaire (surface treatment-independent). long-term quality of life based on the scales of the OHIP questionnaire (surface treatment-independent). The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items. The domain scores can range from 0 to 8. Higher OHIP-14 scores indicate worse and lower scores indicate better OHRQol
Bone resorption measured mesially and distally in millimeters | 36 months
  Determining the long-term difference between different implants in relation to bone erosion around the implant (radiological based on measurements).

CONTACTS AND LOCATIONS:
Overall Officials: Márk Antal, Dr. habil., Principal Investigator — Szeged University
Locations (1):
- SmileDent Kft., Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Derks J, Hakansson J, Wennstrom JL, Tomasi C, Larsson M, Berglundh T. Effectiveness of implant therapy analyzed in a Swedish population: early and late implant loss. J Dent Res. 2015 Mar;94(3 Suppl):44S-51S. doi: 10.1177/0022034514563077. Epub 2014 Dec 11. PMID 25503901
- [Background] van Velzen FJ, Ofec R, Schulten EA, Ten Bruggenkate CM. 10-year survival rate and the incidence of peri-implant disease of 374 titanium dental implants with a SLA surface: a prospective cohort study in 177 fully and partially edentulous patients. Clin Oral Implants Res. 2015 Oct;26(10):1121-8. doi: 10.1111/clr.12499. Epub 2014 Nov 5. PMID 25370914
- [Background] De Angelis F, Papi P, Mencio F, Rosella D, Di Carlo S, Pompa G. Implant survival and success rates in patients with risk factors: results from a long-term retrospective study with a 10 to 18 years follow-up. Eur Rev Med Pharmacol Sci. 2017 Feb;21(3):433-437. PMID 28239830
- [Background] Wang H, Eliaz N, Xiang Z, Hsu HP, Spector M, Hobbs LW. Early bone apposition in vivo on plasma-sprayed and electrochemically deposited hydroxyapatite coatings on titanium alloy. Biomaterials. 2006 Aug;27(23):4192-203. doi: 10.1016/j.biomaterials.2006.03.034. Epub 2006 Apr 18. PMID 16618502
- [Background] Eliaz N, Shmueli S, Shur I, Benayahu D, Aronov D, Rosenman G. The effect of surface treatment on the surface texture and contact angle of electrochemically deposited hydroxyapatite coating and on its interaction with bone-forming cells. Acta Biomater. 2009 Oct;5(8):3178-91. doi: 10.1016/j.actbio.2009.04.005. Epub 2009 Apr 10. PMID 19409870
- [Background] Eliaz N, Ritman-Hertz O, Aronov D, Weinberg E, Shenhar Y, Rosenman G, Weinreb M, Ron E. The effect of surface treatments on the adhesion of electrochemically deposited hydroxyapatite coating to titanium and on its interaction with cells and bacteria. J Mater Sci Mater Med. 2011 Jul;22(7):1741-52. doi: 10.1007/s10856-011-4355-y. Epub 2011 May 25. PMID 21611792
- [Background] Eliaz N, Kopelovitch W, Burstein L, Kobayashi E, Hanawa T. Electrochemical processes of nucleation and growth of calcium phosphate on titanium supported by real-time quartz crystal microbalance measurements and X-ray photoelectron spectroscopy analysis. J Biomed Mater Res A. 2009 Apr;89(1):270-80. doi: 10.1002/jbm.a.32129. PMID 18563813
- [Background] Eliaz N, Eliyahu M. Electrochemical processes of nucleation and growth of hydroxyapatite on titanium supported by real-time electrochemical atomic force microscopy. J Biomed Mater Res A. 2007 Mar 1;80(3):621-34. doi: 10.1002/jbm.a.30944. PMID 17051536
- [Background] Lakstein D, Kopelovitch W, Barkay Z, Bahaa M, Hendel D, Eliaz N. Enhanced osseointegration of grit-blasted, NaOH-treated and electrochemically hydroxyapatite-coated Ti-6Al-4V implants in rabbits. Acta Biomater. 2009 Jul;5(6):2258-69. doi: 10.1016/j.actbio.2009.01.033. Epub 2009 Feb 3. PMID 19251497
- [Background] Fernandez de Grado G, Keller L, Idoux-Gillet Y, Wagner Q, Musset AM, Benkirane-Jessel N, Bornert F, Offner D. Bone substitutes: a review of their characteristics, clinical use, and perspectives for large bone defects management. J Tissue Eng. 2018 Jun 4;9:2041731418776819. doi: 10.1177/2041731418776819. eCollection 2018 Jan-Dec. PMID 29899969
- [Background] Desjardins RP. Hydroxyapatite for alveolar ridge augmentation: indications and problems. J Prosthet Dent. 1985 Sep;54(3):374-83. doi: 10.1016/0022-3913(85)90556-6. PMID 2999379
- [Background] Younes F, Cosyn J, De Bruyckere T, Cleymaet R, Bouckaert E, Eghbali A. A randomized controlled study on the accuracy of free-handed, pilot-drill guided and fully guided implant surgery in partially edentulous patients. J Clin Periodontol. 2018 Jun;45(6):721-732. doi: 10.1111/jcpe.12897. Epub 2018 May 10. PMID 29608793
- [Derived] Antal MA, Kiscsatari R, Braunitzer G, Piffko J, Varga E, Eliaz N. Assessment of a novel electrochemically deposited smart bioactive trabecular coating (SBTC(R)): a randomized controlled clinical trial. Head Face Med. 2024 Apr 16;20(1):24. doi: 10.1186/s13005-024-00426-0. PMID 38627712